CLINICAL TRIAL: NCT00678834
Title: Human Tissue Distribution of Orally Supplemented Natural Vitamin E Tocotrienol
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chandan K Sen (Other)
Collaborators: Carotech Inc. (Industry)
Responsible Party: Sponsor-Investigator, Chandan K Sen, Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2005C0034
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Results first posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-07

CONDITIONS: End Stage Cardiac Failure; Pulmonary Failure; End Stage Liver Disease; Morbid Obesity; Recalcitrant Epilepsy Requiring Surgery; Healthy Subjects
MeSH Terms: conditions — End Stage Liver Disease; Obesity, Morbid | interventions — Tocopherols; Tocotrienols

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Active Comparator): To surgery patients, Tocotrienol capsules. 200mg (2 100mg capsules) to take by mouth twice daily to total 400mg daily
  Interventions: Dietary Supplement: To surgery patients, Tocotrienol capsules.
- Arm 2 (Active Comparator): To surgery patients, Tocopherol capsules. 200mg (2 100mg capsules) to take by mouth twice daily to total 400mg daily
  Interventions: Dietary Supplement: To surgery patients, Tocopherol capsules.
- Arm 3 (Active Comparator): Tocotrienol to healthy subjects - 200 mg to take orally two times a day (400 mg a day).
  Interventions: Dietary Supplement: Tocotrienol to healthy subjects.

INTERVENTIONS:
Dietary Supplement: To surgery patients, Tocopherol capsules. — 200mg (2 100mg capsules) to take by mouth twice daily to total 400mg daily
  Arms: Arm 2
Dietary Supplement: Tocotrienol to healthy subjects. — 200 mg to take orally two times a day (400 mg a day).
  Arms: Arm 3
Dietary Supplement: To surgery patients, Tocotrienol capsules. — 200mg (2 100mg capsules) to take by mouth twice daily to total 400mg daily
  Arms: Arm 1

SUMMARY:
Levels of tocotrienol in human tissues following supplementation is not currently known. The objective of this present study is to determine the levels of this form of vitamin E in the human tissues such as skin, heart, lung, liver, adipose tissue, Brain and cerebrospinal fluid (CSF) following oral supplementation

DETAILED DESCRIPTION:
In nature, there are eight members in the vitamin E family: a-, b-, g- and d-TCP, and a-, b-, g- and d-tocotrienol (TCT). Vitamin E research has developed highly asymmetrically. Out of the 25,000+ papers on vitamin E in the PubMed, 99% deal with tocopherols. Recent research has demonstrated the lack of cancer-preventive effects and potential adverse health consequences of tocopherol (6). As a result, more attention has been turned towards non-tocopherol forms of vitamin E (16). Palm oil represents a major source of natural TCT. TCT possess powerful neuroprotective, antioxidant, anti-cancer and cholesterol lowering properties that often differ from the properties of TCP (15).

During the last five years, our and other laboratories have reported several striking beneficial properties of tocotrienols in experimental settings. One major concern that limits enthusiasm for tocotrienol for humans is the report that the vitamin E transporting protein, tocopherol-transport protein (TTP), has a very low affinity to transport tocotrienol. Using TTP-knock out mice, we have recently demonstrated that oral TCT is effectively carried to vital organs and that such transport can take place independent of TTP. With that background, the purpose of this project is to test the hypothesis that orally supplemented tocotrienol reaches the vital organs of humans.

ELIGIBILITY:
Aim 1 Surgical candidate with a surgery schedule date with a time period of 4-24 weeks (<4 weeks will be excluded; last dose until 24h before surgery) In Aim 1 we expect to have patients, with diverse co-morbidity and medication conditions.

Patient Selection: Because of limitation in obtaining healthy human tissues (as in Aim 2), we plan to obtain these tissues from patients who are scheduled for the following surgeries for subjects in group one:

Heart Heart Transplant Heart Failure- Biopsy taken from diseased heart Lung Lung Transplant, Lung-wedge/resection, Lobectomy Cancer- Tissue sample taken from removed lung or resected portion of lung Liver Liver Transplant, Biopsy, Resection Hepatic Malignancy- Biopsy taken from resected portion of liver Adipose Tissue Panniculectomy Excessive Tissue of the Abdomen Brain & CSF Epilepsy Excised brain tissue and cerebrospinal fluid

To ensure higher enrollment we are not controlling for age of subjects as long as the subjects are 21 years of age or older.

Inclusion Criteria Aim 1:

* age 21 and older
* good health
* non- smoker
* no current medications
* non- pregnant or non-breastfeeding
* no previous use of OTC medications or other form of supplements containing vitamin-E.

Inclusion Criteria Aim 2:

* age 21 - 40 years
* good health
* non- smoker
* no current medications
* non- pregnant or non-breastfeeding
* no previous use of OTC medications or other form of supplements containing vitamin-E.

Exclusion Criteria Aim 1:

* Long-term use of OTC medications containing vitamin-E or current vitamin-E supplements
* Scheduled surgery date lesser than 4 weeks or greater than 24 weeks.

Exclusion Criteria Aim 2:

* Over 40 or under 21 years of age
* Current smoker
* Pregnant and breastfeeding
* Diabetes and HIV diagnosis
* Immunosuppression therapy
* Any neurological problems
* Long-term use of OTC medications containing vitamin-E or current vitamin-E supplements
* ETOH or drug abuse

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandan Sen, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Result] Patel V, Rink C, Gordillo GM, Khanna S, Gnyawali U, Roy S, Shneker B, Ganesh K, Phillips G, More JL, Sarkar A, Kirkpatrick R, Elkhammas EA, Klatte E, Miller M, Firstenberg MS, Chiocca EA, Nesaretnam K, Sen CK. Oral tocotrienols are transported to human tissues and delay the progression of the model for end-stage liver disease score in patients. J Nutr. 2012 Mar;142(3):513-9. doi: 10.3945/jn.111.151902. Epub 2012 Feb 1. PMID 22298568

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1- Surgery + Tocotrienol 200 mg: Surgery Patients to take Tocotrienol capsules.: 200mg (two 100mg capsules) taken by mouth twice to total 400mg daily
- Arm 2- Surgery + Tocopherol 200 mg: Surgery Patients to take Tocopherol capsules.: 200mg (two 100mg capsules) taken by mouth twice to total 400mg daily
- Arm 3- Healthy +Tocotrienol 400 mg: Healthy patients to take Tocotrienol: 400 mg to take orally (two 200 mg capsules) two times a day.
Period: Overall Study
Arm/Group | Arm 1- Surgery + Tocotrienol 200 mg | Arm 2- Surgery + Tocopherol 200 mg | Arm 3- Healthy +Tocotrienol 400 mg
Started | 40 | 15 | 25
Completed | 24 | 15 | 16
Not Completed | 16 | 0 | 9

BASELINE CHARACTERISTICS:
Population: The healthy participants included: age 21-40 y, good health, nonsmoker, nonpregnant or nonbreastfeeding, and no recent (past 6 mo) or current use of supplements containing vitamin E. The surgical participants group included adipose, brain, cardiac muscle, and liver tissue of the surgical participants age 21 and older.
Groups:
- Arm 1- Surgical + Tocotrienol 200 mg: Surgical Subjects will recieve either Tocotrienol: 200mg (two 100mg capsules) to take twice daily by mouth to make a total of 400mg per day
- Arm 2 - Surgical + Tocopherol 200 mg: Surgical Subjects will recieve Tocopherol: 200mg (two 100mg capsules) to take twice daily by mouth to make a total of 400mg per day
- Arm 3- Healthy + Tocotrienol 200 mg: Healthy Subjects will recieve either Tocotrienol: 200mg (two 100mg capsules) to take twice daily by mouth to make a total of 400mg per day
- Total: Total of all reporting groups
Arm/Group | Arm 1- Surgical + Tocotrienol 200 mg | Arm 2 - Surgical + Tocopherol 200 mg | Arm 3- Healthy + Tocotrienol 200 mg | Total
Number analyzed (Participants) | 40 | 15 | 25 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.37 (12.81) | 54 (11.56) | 30.24 (8.59) | 40.37 (4.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 10 | 13 | 43
  Male | 20 | 5 | 12 | 37
Region of Enrollment [Number; unit: participants]
  United States | 40 | 15 | 25 | 80

OUTCOME MEASURES:

1. Primary Outcome: The Levels of TCT in the Tissues of "Non-healthy" Subjects and in the Tissue of "Healthy" Subjects Following Oral Supplementation (200 mg x 2 Per Day for 4-24 Weeks)
Time Frame: After at least 1 month of supplementation
Population: Box plots were used to determine outliers defined as values . the 75th percentile plus 1.5 times the IQR or values , the 25th percentile minus 1.5 times the IQR (20). Outliers were identified and it was determined that laboratory procedural errors were the cause and thus removed from the analysis.
Measure: Mean (Standard Deviation); unit: nmol/g
Groups:
- Arm 1: Surgical, Adipose: adipose aTE levels after supplementation (400mg/d)
- Arm 1: Surgical, Brain: brain aTE levels after supplementation (400mg/d)
- Arm 1: Surgical, Heart: heart aTE levels after supplementation (400mg/d)
- Arm 1: Surgical, Liver: liver aTE levels after supplementation (400mg/d)
- Arm 2: Surgical, Adipose: adipose aTCP levels after supplementation (400mg/d)
- Arm 2: Surgical, Brain: brain aTCP levels after supplementation (400mg/d)
- Arm 2: Surgical, Heart: heart aTCP levels after supplementation (400mg/d)
- Arm 2: Surgical, Liver: liver aTCP levels after supplementation (400mg/d)
- Arm 3: Healthy, Blood, Week 0: Baseline blood levels of aTE prior to supplementation
- Arm 3: Healthy, Blood, Week 6: Blood levels of aTE after 6 weeks of supplementation (400mg/d)
- Arm 3: Healthy, Skin, Week 12: skin levels of aTE after 12 weeks of supplementation (400mg/d)
- Arm 3: Healthy, Skin, Week 0: baseline skin levels of aTE prior to supplementation
- Arm 3: Healthy, Blood, Week 12: Blood levels of aTE after 12 weeks of supplementation (400mg/d)
Arm/Group | Arm 1: Surgical, Adipose | Arm 1: Surgical, Brain | Arm 1: Surgical, Heart | Arm 1: Surgical, Liver | Arm 2: Surgical, Adipose | Arm 2: Surgical, Brain | Arm 2: Surgical, Heart | Arm 2: Surgical, Liver | Arm 3: Healthy, Blood, Week 0 | Arm 3: Healthy, Blood, Week 6 | Arm 3: Healthy, Skin, Week 12 | Arm 3: Healthy, Skin, Week 0 | Arm 3: Healthy, Blood, Week 12
Number analyzed (Participants) | 5 | 4 | 5 | 4 | 4 | 4 | 3 | 3 | 16 | 16 | 16 | 16 | 16
nmol/g | 9.94 (6.9) | 1.29 (1.06) | 5.37 (4.28) | 0.42 (0.43) | 28.6 (20.7) | 50.5 (17.2) | 31.9 (20.0) | 64.3 (14.9) | 0.01 (0.02) | 1.9 (0.7) | 1.5 (1.8) | 2.5 (3.0) | 0.03 (0.1)

ADVERSE EVENTS:
Groups:
- Arm 1: Surgery patients to take Tocotrienol capsules.: 200mg (two 100mg capsules)taken by mouth twice with foold to make a total of 400mg daily
- Arm 2: Surgery patients to take Tocopherol capsules.: 200mg (two 100mg capsules)taken by mouth twice with foold to make a total of 400mg daily
- Arm 3: Healthy patients to take either Tocotrienol or Tocopherol: 200mg (two 100mg capsules)taken by mouth twice with foold to make a total of 400mg daily
Arm/Group | Arm 1 | Arm 2 | Arm 3
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/15 | 0/25
Other Adverse Events (participants affected / at risk) | 0/40 | 0/15 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No